CLINICAL TRIAL: NCT06169982
Title: A Phase 1, Open-Label, Multiple-Dose Study to Investigate Steady-State Pharmacokinetics and Pharmacodynamics During a Euglycemic Clamp of LY3209590 in Participants With Type 2 Diabetes Mellitus
Brief Title: A Multiple Dose Study of LY3209590 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18811; I8H-MC-BDDG (Other: Eli Lilly and Company); 2023-508008-39-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Clamp; Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3209590 (Experimental): LY3209590 administered subcutaneously (SC)
  Interventions: Drug: LY3209590

INTERVENTIONS:
Drug: LY3209590 — Administered SC

SUMMARY:
The purpose of this study is to measure the activity and insulin time action of LY3209590 at steady state in participants with type 2 diabetes mellitus. The total study duration is approximately 182 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 2 Diabetes (T2DM).
* Participants who are insulin naive or receiving basal insulin [NPH (neutral protamine Hagedorn) once or twice daily, once-daily insulin glargine U100 or U300, once-daily insulin degludec, or insulin detemir once or twice daily] for fewer than 5 years prior to screening.
* Have glycated hemoglobin (HbA1c) of ≥7.0 percent (%) to ≤9.5%, HbA1c of ≥6.5% to ≤9.5% for participants on treatment with sulfonylureas and/or Sodium-Glucose Transport Protein 2 inhibitors who require washout.
* Have a body mass index between 27 and 40 kilograms per meter square.
* Male or female participants who are willing to comply with the contraception requirements consistent with local regulations.
* Be willing to allow blood sample collection, reliable and to be available for the duration of the study as required for the study protocol.

Exclusion Criteria:

* Have known or suspected allergic reactions to study drugs, related compounds, excipients, and devices used in the study.
* Have a specific type of diabetes other than T2DM.
* Have known hemoglobinopathy, hemolytic anemia or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the measurement of HbA1c.
* Participants with a history of kidney complications.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the concentration curve during one dosing interval at steady state (AUCss) of LY3209590 | One dosing interval at steady state from 0 to 168 hours after last dose
  PK: AUCss of LY3209590

SECONDARY OUTCOMES:
PK: Total amount of glucose infused during one dosing interval at steady state (Gtot,SS) of LY3209590 | One dosing interval at steady state from 0 to 168 hours after last dose
  PK: Gtot,SS of LY3209590

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No